CLINICAL TRIAL: NCT00679146
Title: Efficacy and Safety of a Fixed Combination (Thiocolchicoside 8 mg + Ketoprofen 100 mg ) Compared to Thiocolchicoside 8 mg Administered Twice a Day for 7 Days in Patients Suffering From Acute Non Specific Low Back Pain
Brief Title: Efficacy Safety of a Combination Thiocolchicoside+Ketoprofen Compared to Thiocolchicoside Twice a Day for 7 Days in Patients Suffering From Acute Non Specific Low Back Pain
Acronym: TIOKET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, Sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KETOP_R_02693
Record Dates: First submitted 2008-05-06; First posted 2008-05-16 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — thiocolchicoside

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): 1 tablet TCC 8 mg + ketoprofen 100 mg b.i.d + 2 tablets TCC placebo b.i.d
  Interventions: Drug: Thiocolchicoside+Ketoprofen
- 2 (Active Comparator): 2 tablets TCC 4 mg b.i.d. + 1 tablet of FDC placebo b.i.d
  Interventions: Drug: Thiocolchicoside

INTERVENTIONS:
Drug: Thiocolchicoside+Ketoprofen — 1 tablet TCC 8 mg + ketoprofen 100 mg b.i.d + 2 tablets TCC placebo b.i.d
  Arms: 1
Drug: Thiocolchicoside — 2 tablets TCC 4 mg b.i.d. + 1 tablet of FDC placebo b.i.d
  Arms: 2

SUMMARY:
Primary Objective :

To demonstrate the superiority of the oral fixed - combination of a muscle relaxant, thiocolchicoside (TCC) to a non steroidal anti-inflammatory drug, ketoprofen, over oral TCC, on average pain within the last 24 hours in adults suffering from acute non specific low back pain with an episode of recent onset

Secondary Objective :

To compare the safety of the oral combination to that of oral TCC alone

ELIGIBILITY:
List of Inclusion and Exclusion criteria :

Inclusion Criteria:

* Non specific low back pain with an acute episode of recent onset (<48 hours) defined by average pain within the last 24 hours equal or more than 50 mm on the Visual Analogue Scale (VAS)
* Low back pain of diagnosis category 1 (low back pain radiating no farther than the intergluteal fold) or 2 (low back pain radiating no farther than the knee), as defined by the International Paris Task Force on Back Pain

Exclusion Criteria:

Exclusion criteria related to study methodology:

* Low back pain due to vertebral collapse or of no mechanical origin (suspected by history taking and physical examination), such as neoplasm, infection or inflammatory disorders,
* Low back pain of diagnosis category 3 (low back pain radiating beyond the knee, with no neurologic signs) or 4 (low back pain radiating to a precise and entire leg dermatome, with or without neurologic signs), as defined by the International Paris Task Force on Back Pain
* History of inflammatory arthritis of large joints,
* History of seizure disorders,
* History of malignant tumour,
* Treatment with steroidal agents (including aspirin) during the two days prior to prospective inclusion, prolonged used of corticosteroids,
* Treatment with NSAIDs or muscle relaxant or opioid analgesics within 3 days of admission,
* Psychiatric or mental diseases,
* Immunosuppression, HIV,
* Inclusion in another study in the past six months or previous inclusion in this study,
* History of alcohol, drugs or narcotics abuse
* Recent history of violent trauma,
* Constant progressive, non mechanical pain (no relief with bed rest),
* Thoracic pain,
* Patient systemically unwell,
* Unexplained weight loss,
* Widespread neurological symptoms (including cauda equine syndrome),
* Structural deformity
* Fever,
* Clinical significant renal dysfunction defined by Creatinine > 1.5 UNL,
* Clinically significant hepatic dysfunction defined by:
* Total Bilirubin > 2 UNL
* SGOT (AST) > 1.5 UNL
* SGPT (ALAT) > 1.5 UNL
* Alkaline Phosphatase > 1.5 UNL
* Patients who have received other therapy (physiotherapy, physical manipulations, invasive intervention, acupuncture therapy...) within the last 48 hours.

Exclusion criteria related to trial drugs:

* Pregnancy, breast feeding or women of childbearing potential not using efficient contraception. Patient with Intra Uterine Device should use another form of contraception as the efficacy of the IUD may be reduced by ketoprofen.

Exclusion criteria related to thiocolchicoside:

* Known or suspected hypersensitivity to thiocolchicoside

Exclusion criteria related to ketoprofen:

* Uncontrolled heart failure,
* Arterial Hypertension (SBP>140 mmHg or DBP >90 mmHg),
* Stroke or myocardial infarction in the past,
* Myopathy
* Myasthenia,
* History of active peptic ulcer or gastrointestinal (GI) bleeding, history of gastric pain with NSAIDs,
* History of NSAID/aspirin-induced asthma,
* Known or suspected hypersensitivity to ketoprofen.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 334 (Actual)
Dates: Start 2008-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Average pain within the last 24 hours (VAS) | at D3 visit

SECONDARY OUTCOMES:
Average pain within the last 24 hours (VAS) | at D7 visit

CONTACTS AND LOCATIONS:
Overall Officials: Margarita MURRIETA-AGUTTES, Study Director — Sanofi
Locations (6):
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Bogotá, Colombia
- Sanofi-Aventis Administrative Office, Cairo, Egypt
- Sanofi-Aventis Administrative Office, Guatemala City, Guatemala
- Sanofi-Aventis Administrative Office, Col. Coyoacan, Mexico
- Sanofi-Aventis Administrative Office, Caracas, Venezuela